CLINICAL TRIAL: NCT04388644
Title: Department of Chinese Medicine, Branch of Linsen, Chinese Medicine, and Kunming, Taipei City Hospital, Taipei, Taiwan Institute of Traditional Medicine, National Yang-Ming University, Taipei, Taiwan.
Brief Title: Survey of Satisfaction on Traditional Chinese Medicine Jing-Guan-Fang (JGF) for COVID-19 Prevention
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei City Hospital (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Other Study IDs: TCHIRB-10904015-E
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-02

CONDITIONS: Corona Virus Infection
Keywords: natural herbal medicine; Chinese medicine
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the retrospective observation study, the first line to care CAVID-19

DETAILED DESCRIPTION:
The satisfaction of using nature herbal medicine for frontline medical staffs to prevent COVID-19: a retrospective clinical study.

The medical frontline staffs have the high risk to be infected during working. The stress and load were acuminated, especially when they got the similar symptoms as COVID-19. NHM has been used to early prevention for thousands of years9-12. It was well accept to take NHM for early prevention in many Asia-Pacific countries. Although many NHM remedies of COVID-19 treatment or prevention were reported, but the related study were lacking. To understand the pressure and the satisfaction of frontline medical staffs after taking JGF for early prevention we conducted this retrospective clinical study to explore the relationship in different groups.

ELIGIBILITY:
Inclusion Criteria:

* The person first-line medical staff in hospital
* the inspection personnel in airport
* self-quarantine at home.
* self-quarantine at office.

Exclusion Criteria:

* no willing to participate
* allergy to herbal medicine
* severe illness evaluated by physician

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The first-line medical staff who take care of COVID-19 patients in public hospital northern Taiwan., and the self-quarantine who have contacted with history.
  Some of the population will take natural herbal medicine to prevent COVID-19 infection.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-05-20 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
the number confirmed COVID-19 cases | 8 weeks
  The isolated person and first-line care person who taking JGF
The person with COVID-19 like symptoms | 8 weeks
  The isolated person and first-line care person who taking JGF

SECONDARY OUTCOMES:
The improving rate of COVID-19 like symptoms | 8 weeks
  The isolated person and first-line care person who taking JGF
The satisfaction% to taking JGF | 8 weeks
  The isolated person and first-line care person who taking JGF

CONTACTS AND LOCATIONS:
Overall Officials: Chung-HUa Hsu, PhD, Study Director — Taipei City Hospital
Locations (3):
- Taiwan (3):
  - Branch of Chinese Medicine, Taipei City Hospital, Taipei
  - Branch of Linsen Chinese Medicine and Kunming, Taipei City Hospital, Taipei
  - Taipei City Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No